CLINICAL TRIAL: NCT06008769
Title: Cognitive-Behavioral Therapy for Opioid Use Disorder: A Manualized Pilot Study
Brief Title: Therapy for People With Opioid Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia College of Osteopathic Medicine (Other)
Collaborators: Prevention Point Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H23-025
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 Week Manualized Cognitive-Behavioral Therapy Intervention (Experimental): Participants will receive a once-per-week, 12 week manualized cognitive-behavioral therapy intervention.
  Interventions: Behavioral: 12 Week Manualized Cognitive-Behavioral Therapy Intervention

INTERVENTIONS:
Behavioral: 12 Week Manualized Cognitive-Behavioral Therapy Intervention — The manualized intervention, Cognitive Behavioral Therapy for Opioid Use Disorder, was co-written and developed by the study PI, Dr. Lent (see Appendix). The manual consists of one module (Module 0) on assessment and 12 modules of CBT. This study will focus on delivery of Modules 1-12 that focus on several tenets of CBT, including skill development (cognitive restructuring, refusal skills, problem-solving, coping strategies), functional analysis (triggers, reinforcement) and utilizing the cognitive model.

SUMMARY:
The goal of this pilot clinical trial is to test the feasibility of a 12-week manualized cognitive-behavioral therapy treatment for opioid use disorder in reducing or stopping illicit opioid use in a community setting. Participants will complete 12 weeks of therapy with a behavioral health counselor and will complete assessments at baseline and 12 weeks. Other outcomes include changes in mood and perceptions of recovery-related support after 12 weeks of therapy.

DETAILED DESCRIPTION:
Cognitive-Behavioral Therapy (CBT) is one of the most well-supported and widely used psychosocial treatments for substance use disorders (SUDs); however, few studies have evaluated the efficacy of CBT for opioid use disorder (OUD). This prospective, longitudinal pilot study (pre-post design) will assess the feasibility of the first manualized CBT treatment for OUD in adults (N = 20) in a community-based setting (Prevention Point Philadelphia). This study will utilize clinical (urinalysis), patient-reported, and provider-reported outcomes (mood, support, feasibility, satisfaction with treatment) over 12 weeks of a manualized cognitive-behavioral treatment for OUD. This prospective, longitudinal pilot study will evaluate the feasibility of a novel psychotherapy for OUD. This study will utilize both clinical (urinalysis) and patient or provider-reported (mood, support, feasibility) outcomes to assess the feasibility of 12 weeks of manualized cognitive-behavioral treatment for OUD. All study recruitment, consent and intervention delivery will occur at Prevention Point (2913-15 Kensington Ave, Philadelphia, PA). Outcomes will include participant-reported treatment satisfaction, as well as EMR-extracted clinical data (session attendance, urinalysis, mood, demographics, medical information, and recovery-related support).

We hypothesize that individuals with OUD will demonstrate a reduction illicit opioid use from baseline to week 12 as assessed by urinalysis (% change, positive/negative). As a secondary outcome, use of other substances will also be assessed from baseline to week 12 (e.g., alcohol, cocaine). Use of medication for OUD (MOUD; e.g., buprenorphine. methadone) will be accounted for in analyses.

We hypothesize that mood and perceptions of recovery-related resources will improve from baseline to week 12.

As an exploratory aim, we will evaluate intervention feasibility through electronic medical record (EMR) data of number of sessions attended over 12 weeks, treatment fidelity checklists, and a participant survey of treatment satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patient at Prevention Point Philadelphia
* 18 years or older
* Living with opioid use disorder
* Has a goal to reduce or eliminate illicit opioid use
* Able to provide informed consent

Exclusion Criteria:

* Not comfortable receiving psychotherapy in English
* Under custodial supervision through the legal justice system (e.g., halfway house following incarceration, involuntary detention or confinement, status as a "prisoner")

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-08-06 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Urinalysis-confirmed Reduction or Elimination of Illicit Opioid Use | Baseline, 12 weeks

SECONDARY OUTCOMES:
The Patient Health Questionnaire-9 (PHQ-9) | Baseline, 12 weeks
  The PHQ-9 is a nine-item instrument (0-3 Likert type scale) for monitoring and measuring depression severity over the past two weeks. The PHQ-9 has strong validity and reliability and is frequently used in clinical settings. The PHQ-9 is scored on a 4-point Likert-type scale, with the lowest value being "Not at All" and the highest value being "Nearly Every Day" with higher overall scores indicating more severe depression.
The Brief Assessment of Recovery Capital (BARC-10) | Baseline, 12 weeks
  The BARC-10 is a 10-item measure assessing the perceived characteristics and assets and individual develops on their recovery journey. The BARC-10 has high internal consistency (α = .90). The BARC-10 is scored on a 6-point Likert-type scale ranging from "Strongly Disagree" to "Strongly Agree" with higher scores indicating higher recovery capital.
The Client Satisfaction Questionnaire-8 (CSQ-8) | 12 weeks
  The CSQ-8 is a brief, eight-item treatment satisfaction questionnaire. The CSQ-8 is scored on a series of 4-point Likert-type scales, with higher scores indicating greater treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Lent, PhD, Principal Investigator — Philadelphia College of Osteopathic Medicine
Locations (1):
- Prevention Point Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kampman K, Jarvis M. American Society of Addiction Medicine (ASAM) National Practice Guideline for the Use of Medications in the Treatment of Addiction Involving Opioid Use. J Addict Med. 2015 Sep-Oct;9(5):358-67. doi: 10.1097/ADM.0000000000000166. PMID 26406300
- [Background] Center for Substance Abuse Treatment. Clinical Guidelines for the Use of Buprenorphine in the Treatment of Opioid Addiction. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2004. Report No.: (SMA) 04-3939. Available from http://www.ncbi.nlm.nih.gov/books/NBK64245/ PMID 22514846
- [Background] Guidelines for the Psychosocially Assisted Pharmacological Treatment of Opioid Dependence. Geneva: World Health Organization; 2009. Available from http://www.ncbi.nlm.nih.gov/books/NBK143185/ PMID 23762965
- [Background] Dugosh K, Abraham A, Seymour B, McLoyd K, Chalk M, Festinger D. A Systematic Review on the Use of Psychosocial Interventions in Conjunction With Medications for the Treatment of Opioid Addiction. J Addict Med. 2016 Mar-Apr;10(2):93-103. doi: 10.1097/ADM.0000000000000193. PMID 26808307
- [Background] Seth P, Scholl L, Rudd RA, Bacon S. Overdose Deaths Involving Opioids, Cocaine, and Psychostimulants - United States, 2015-2016. MMWR Morb Mortal Wkly Rep. 2018 Mar 30;67(12):349-358. doi: 10.15585/mmwr.mm6712a1. PMID 29596405
- [Background] McHugh RK, Hearon BA, Otto MW. Cognitive behavioral therapy for substance use disorders. Psychiatr Clin North Am. 2010 Sep;33(3):511-25. doi: 10.1016/j.psc.2010.04.012. PMID 20599130
- [Background] Substance Abuse and Mental Health Services Administration. Behavioral health treatments and services; 2017. Retrieved from https://www.samhsa.gov/treatment. Accessed September 6. 2018.
- [Background] Beck AT. Cognitive therapy: nature and relation to behavior therapy. Behav Ther. 1970;1(2),184-200.
- [Background] Ellis A. Reason and Emotion in Psychotherapy. New York, NY: Stuart; 1962.
- [Background] Festinger DS, Lent MR. Cognitive-Behavioral Therapy (CBT) for the Treatment of Opioid Use Disorder. Trafford Publishing; 2022 Aug 18.
- [Background] Lent MR, Callahan HR, Womer P, Mullen PM, Shook CB, DiTomasso RA, Felgoise SH, Festinger DS. A mental health professional survey of cognitive-behavioral therapy for the treatment of opioid use disorder. J Clin Psychol. 2021 Jul;77(7):1607-1613. doi: 10.1002/jclp.23170. Epub 2021 May 10. PMID 33971028
- [Background] Moore BA, Barry DT, Sullivan LE, O'connor PG, Cutter CJ, Schottenfeld RS, Fiellin DA. Counseling and directly observed medication for primary care buprenorphine maintenance: a pilot study. J Addict Med. 2012 Sep;6(3):205-11. doi: 10.1097/ADM.0b013e3182596492. PMID 22614936
- [Background] Fiellin DA, Barry DT, Sullivan LE, Cutter CJ, Moore BA, O'Connor PG, Schottenfeld RS. A randomized trial of cognitive behavioral therapy in primary care-based buprenorphine. Am J Med. 2013 Jan;126(1):74.e11-7. doi: 10.1016/j.amjmed.2012.07.005. PMID 23260506
- [Background] Ling W, Hillhouse M, Ang A, Jenkins J, Fahey J. Comparison of behavioral treatment conditions in buprenorphine maintenance. Addiction. 2013 Oct;108(10):1788-98. doi: 10.1111/add.12266. Epub 2013 Jul 12. PMID 23734858
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Gilbody S, Richards D, Brealey S, Hewitt C. Screening for depression in medical settings with the Patient Health Questionnaire (PHQ): a diagnostic meta-analysis. J Gen Intern Med. 2007 Nov;22(11):1596-602. doi: 10.1007/s11606-007-0333-y. Epub 2007 Sep 14. PMID 17874169
- [Background] Vilsaint CL, Kelly JF, Bergman BG, Groshkova T, Best D, White W. Development and validation of a Brief Assessment of Recovery Capital (BARC-10) for alcohol and drug use disorder. Drug Alcohol Depend. 2017 Aug 1;177:71-76. doi: 10.1016/j.drugalcdep.2017.03.022. Epub 2017 May 19. PMID 28578224